CLINICAL TRIAL: NCT02064114
Title: Supervised Obesity Reduction Trial for AF Ablation Patients
Brief Title: SORT - AF Supervised Obesity Reduction Trial for AF Ablation Patients
Acronym: SORT-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Abbott Medical Devices (Industry); Deutsches Zentrum für Herz-Kreislauf-Forschung (DZHK) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PV4300
Record Dates: First submitted 2014-02-13; First posted 2014-02-17 (Estimated); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Atrial Fibrillation; Obesity; Sleep Apnea
Keywords: BMI >40
MeSH Terms: conditions — Atrial Fibrillation; Obesity; Sleep Apnea Syndromes | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Active Comparator): Start of optimal management of risk factors, every 2 weeks for 6 months after atrial fibrillation ablation. And followed for a period of 3,6 and 12 months after the procedure.
  Interventions: Procedure: Intervention group
- control group (Active Comparator): conventional treatment, followed for a period of 3,6 and 12 months after the procedure.
  Interventions: Procedure: control group

INTERVENTIONS:
Procedure: Intervention group — Start of optimal management of risk factors, every 2 weeks for 6 months after atrial fibrillation ablation. And followed for a period of 3,6 and 12 months after the procedure.
  Arms: Intervention group
Procedure: control group — Followed for a period of 3,6 and 12 months after the procedure.
  Arms: control group

SUMMARY:
Study hypothesis:

Weight reduction in obese patients with atrial fibrillation. Obese patients benefit from an obesity treatment after atrial fibrillation ablation.

Study design:

A prospective randomized, open-label clinical trial.

DETAILED DESCRIPTION:
Study protocol:

The purpose of this study is to proof a professional care of overweight patients with symptomatic atrial fibrillation, as well as the treatment of the risk factors for atrial fibrillation, especially obstructive sleep apnea and hypertension.

There is a 1:1 randomization. In the intervention group, patients are followed up in a 6-month intensive care after atrial fibrillation ablation. During the follow up time patients will visit the nutritional advice every two weeks for 6 months.

The Follow-up in the control group is standard of care. At baseline, a screening test for obstructive sleep apnea and arterial hypertension will be performed as standard care.

The documentation of atrial fibrillation after ablation is made possible by the implantation of an event recorder before atrial fibrillation ablation.

Follow up:

A follow-up will be performed after 3,6 and 12 months in both groups. Patients in the intervention group will be followed-up every 2 weeks in the first 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Overweight with a BMI ≥ 30
* Obtained written informed consent
* Symptomatic atrial fibrillation with indication for ablation

Exclusion Criteria:

* Age <18 years
* Permanent atrial fibrillation (failed Cardioversion or episode duration > 12 months)
* Previous surgical or interventional therapy of atrial fibrillation
* BMI > 40
* Pregnant women or women of childbearing potential without a negative pregnancy test within 48 hours prior to treatment
* History of hemorrhagic diathesis or other coagulopathies
* Contraindications for oral anticoagulation
* Hyper- or hypothyroidism
* Drug or chronic alcohol abuse
* Has any condition that would make participation not be in the best interest of the subject
* Incompliance
* Unable to perform athletic exercise due to disease or disability
* Resident outside Hamburg

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2020-01-16 (Actual); Study Completion 2020-01-16 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of the study is defined as AF burden between 3 to 12 months after first AF ablation | 12 months
  AF burden is defined as overall percentage of AF during the observed period.

SECONDARY OUTCOMES:
AF burden between 0 and 12 months after first AF ablation | 12 months
AF burden between 0 and 3, 3 to 6 and 6 to 12 months after first AF ablation | 12 months
Freedom of AF (after 3 months blanking period) | 12 months
Time to first recurrent AF (after 3 months blanking period) | 12 months
Body Mass Index (BMI) change from BL to 12 months | 12 months
Exercise capacity change from BL to 12 months | 12 months
Mean blood pressure change from BL to 12 months | 12 months
Number of repeated AF ablation procedures | 12 months
Antiarrhythmic drug therapy at 12 months Antiarrhythmic drug therapy at 12 months Antiarrhythmic drug therapy at 12 months | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Christian Meyer, Principal Investigator — University Heart Center Hamburg
Locations (4):
- Germany (4):
  - Universitäres Herzzentrum Lübeck, Lübeck, Schleswig-Holstein
  - Herzzentrum der Universität zu Köln, Cologne
  - Asklepios ST. Georg, Hamburg
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gessler N, Willems S, Steven D, Aberle J, Akbulak RO, Gosau N, Hoffmann BA, Meyer C, Sultan A, Tilz R, Vogler J, Wohlmuth P, Scholz S, Gunawardene MA, Eickholt C, Luker J. Supervised Obesity Reduction Trial for AF ablation patients: results from the SORT-AF trial. Europace. 2021 Oct 9;23(10):1548-1558. doi: 10.1093/europace/euab122. PMID 33895833